CLINICAL TRIAL: NCT02570438
Title: Improving Surgical Safety of Seniors Through Preoperative Cognitive Screening
Status: Terminated | Type: Observational
Why Stopped: This study was terminated prior to its planned enrollment due to low recruitment rates at the time that the funding for the study was completed.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Newton-Wellesley Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gregory J. Crosby, M.D., Physician, Brigham and Women's Hospital
Other Study IDs: 2015P001020
Record Dates: First submitted 2015-09-30; First posted 2015-10-07 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Cognitive Impairment
Keywords: postoperative outcomes; older surgical patients
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older surgical patients: older patients (≥ 65 years of age) presenting to Massachusetts General Hospital (MGH) or Newton-Wellesley Hospital (NWH) for elective noncardiac, non-neurological surgery requiring hospital admission

SUMMARY:
The hypothesis is that structured preoperative cognitive screening of seniors is feasible without specialized staff and can help preoperatively identify persons at high risk of complications. To demonstrate generalizability of the single center experience, and strengthen the case for routine preoperative cognitive screening of seniors, the aims of this proposal are to implement preoperative cognitive screening of seniors in the preoperative clinics of a community hospital (NWH) and a 2nd tertiary care institution (MGH); and determine whether impairment is an independent predictor of adverse perioperative events.

DETAILED DESCRIPTION:
The overriding hypothesis is that structured preoperative cognitive screening of seniors is feasible without specialized staff and can help preoperatively identify persons at high risk of complications. To demonstrate generalizability of the single center experience, and strengthen the case for routine preoperative cognitive screening of seniors, the aims of this proposal are to implement preoperative cognitive screening of seniors in the preoperative clinics of a community hospital (NWH) and a 2nd tertiary care institution (MGH); and determine whether impairment is an independent predictor of adverse perioperative events. We will enroll seniors (≥ 65 years of age) presenting to Massachusetts General Hospital (MGH) or Newton-Wellesley Hospital (NWH) for elective noncardiac, non-neurological surgery requiring hospital admission (N = 250 each). Study staff will be deployed to one of the sites each day according to a randomization scheme to avoid bias (thus, at each site, recruitment will on average occur 10 d per month). A study team member will obtain informed consent if the patient agrees to participate and satisfies eligibility criteria. Exclusion criteria will be planned ICU admission postoperatively; history of stroke or brain tumor; uncorrected vision or hearing impairment (unable to see pictures or read or hear instructions); limited use of the dominant hand (limited ability to draw); and/or inability to speak, read or understand English.Study staff will use the computerized scheduling system, which is updated continuously in real time and captures relevant information such as age and procedure, to identify potential subjects. When patients check in with the receptionist for their appointment they will be notified that they may be eligible to participate in a study in the CPE involving patients over the age of 65. The receptionist will then provide them with a brochure about the study that includes information about the purpose of the study, the risks to the patient, and the potential benefits to society. The patient will then be asked if they are willing to speak with one of the study investigators and only those patients that agree to speak with a study investigator will be approached. The staff member will then describe the goals and risks of the study in a quiet room and ask the patient if they choose to participate. After all questions have been answered and the patient has the opportunity to read the consent form, written consent will be obtained by one of the study investigators. After obtaining informed consent, the interviewer will ask the patient and informant (if available) "Have you spoken to your doctor about or been evaluated for a change in memory or thinking?" Study staff will also gather a variety of demographic, functional, and medical information by direct questioning and review of the medical record. Specifically, we will collect data on age, years of education, living situation, history of falls, ASA physical status, metabolic equivalents (METS), medication history, and Charlson Comorbidity index. We will administer standard instruments to assess mood (Geriatric Depression Scale-Short [GDS], a 15-item self-report questionnaire, and health and functional status (basic and instrumental activities of daily living [ADLs and IADLs, respectively, and the SF36]), and measure grip strength with a Jamar hand dynamometer as an index of frailty.The SF36 survey profiles physical and mental health and quality-of-life. In addition, it will take one-minute to administer the Animal Fluency Test. This is a cognitive screen that has been shown to be useful in identifying patients at risk of developing postoperative delirium. The World Health Organization Disability Assessment Schedule 2.0 will also be administered as a potential alternative to the SF36 in measuring physical health and disability. Each enrolled patient will also receive a business card listing the investigators' contact information and be advised to expect a follow up telephone call 6 months after surgery to verify data elements and reassess functional outcome.The MiniCog will be used for preoperative cognitive screening. Preoperative clinic staff will perform and score the MiniCog during the preoperative visit, and a study staff member will independently score each test subsequently. The MiniCog involves 3-item recall for memory and a clock drawing test that serves as a distractor. The MiniCog tests visuospatial representation, recall, and executive function. The MiniCog takes just 2-4 min to complete but has been validated in community-based populations, has minimal education, language, or ethnic bias, high sensitivity and specificity for impaired cognition, and age-adjusted normative data are available. Moreover, the pilot data at BWH show the MiniCog is well accepted by geriatric surgical patients, is easy for caregivers of different types to administer and score, and has high inter-rater reliability in a preoperative clinic setting. Probable cognitive impairment will be defined as a MiniCog score ≤ 2 (out of 5) but ordinal scores will also be considered in the data analysis. A score ≤ 2 is a standard cutoff and has ~75% sensitivity and ~90% or greater specificity for MCI or dementia when compared to longer screening and assessment instruments.

Primary outcome measures for feasibility (Aim 1) will be rate of successful testing (a score-able test) and accuracy of scoring (vs. an investigator). Secondary feasibility outcome measures will be perspective of the practitioner about cognitive screening (survey of MGH and NWH CPE staff) and the impact of testing on patient flow at each institution. The latter will be obtained by extracting and comparing data from the CPE's computerized patient flow tracking system on time spent with a provider in a preoperative evaluation room and total duration of the CPE visit (check-in time to departure time) between enrolled subjects and age and procedure matched patients seen in the CPE the previous year. The primary patient outcomes (Aim 2) will be delirium, discharge to a place other than home, and functional outcome (change in SF36); secondary outcomes will be hospital length of stay (LOS), complications (including in-hospital falls), and 30 d readmission rate or mortality. Delirium will be assessed directly on postoperative days 1, 2, and 3 by a member of the study team using the Confusion Assessment Method (CAM), a well-validated measure of delirium in surgical patients.The remaining outcomes data will be extracted from the medical record or electronic databases. Both institutions track time spent in the CPE (with provider, in the lab, in the waiting room, etc.) and have databases that tabulate numerous elements of the hospital event such as age, gender, and race, surgical service, procedure, DRG codes, admit and discharge dates (LOS), and discharge disposition (home, home with services, rehabilitation, skilled nursing facility).

ELIGIBILITY:
Inclusion Criteria:

* patients 65 years of age or older
* presenting to Massachusetts General Hospital (MGH) or Newton-Wellesley Hospital (NWH)
* scheduled for elective noncardiac, non-neurological surgery requiring hospital admission

Exclusion Criteria:

* planned ICU admission postoperatively
* history of stroke or brain tumor
* uncorrected vision or hearing impairment
* limited use of the dominant hand
* inability to speak, read or understand English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: patients 65 years of age or older presenting to Massachusetts General Hospital (MGH) or Newton-Wellesley Hospital (NWH) for elective noncardiac, non-neurological surgery requiring hospital admission. Exclusion criteria will be planned ICU admission postoperatively; history of stroke or brain tumor; uncorrected vision or hearing impairment (unable to see pictures or read or hear instructions); limited use of the dominant hand (limited ability to draw); and/or inability to speak, read or understand English.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
CAM score postoperative days 1-3 | up to 3 days after surgery
  patient score on the confusion assessment method on postoperative day 1, 2, and 3

SECONDARY OUTCOMES:
Discharge location (defined home vs. other than home) on day of discharge from hospital | up to 1 month from the date of surgery
  discharge location (home vs. other than home) will be recorded on the day the patient is discharged from the hospital
Number of newly diagnosed health complications following surgery | up to 30 days after surgery
  number of newly diagnosted health complications up to 30 days after surgery including: Myocardial Infarction, CHF, Cardiac Arrest, Arrythmia, Pneumonia, PE, Reintubation, Stroke, Delirium, Coma>24h, Postoperative deep wound infection, Superficial wound infection, Sepsis, Renal Failure, UTI, Reoperation, DVT, ICU admission
30 day readmission to the hospital or admission to the emergency room | 30 days post surgery
  a patient's readmission to the hospital or admission to the emergency room
30 day mortality | 30 days post surgical procedure
  Patient mortality within 30 days after the surgical procedure
6-month functional health assessment | 6 months post surgical procedure
  Follow up health assessment using the the SF36 or the World Health Organization Disability Assessment Schedule 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Culley, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: No